CLINICAL TRIAL: NCT04803357
Title: A Study on the Use of Real -Time Continuous Glucose Monitoring (RT-CGM) in Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Nicole Ehrhardt, Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00011755
Record Dates: First submitted 2020-11-29; First posted 2021-03-17 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Real- time continuous glucose monitoring using the DexCom G6.
Masking Description: If you are in the control group, you will not be given a RT-CGM. Instead, you will be given a blinded CGM device. You will not be able to view your blood sugar results on the blinded CGM device. If you are in the control group, you will also be given a blood glucose meter to check your glucose using finger sticks according to the recommendations of your provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control : Blinded Continuous Glucose Monitoring (CGM) (No Intervention): If you are in the control group, you will wear a continuous glucose monitor but it will be blinded during pregnancy.
- Intervention: Real Time -Continuous Glucose Monitoring (RT-CGM) (Active Comparator): Wearing RT- CGM during pregnancy
  Interventions: Device: Continuous glucose monitor

INTERVENTIONS:
Device: Continuous glucose monitor — We are offering you an opportunity to wear a medical device that monitors your blood sugars (glucose). This device is called a continuous glucose monitor (CGM). The CGM measures glucose levels through a tiny plastic filament that is inserted under the skin in your abdomen by a skin prick. Typically, you cannot feel this device once it is inserted.
  Arms: Intervention: Real Time -Continuous Glucose Monitoring (RT-CGM)

SUMMARY:
The purpose of this study is to examine whether RT-CGM (real time continuous glucose monitoring) use improves glucose control, maternal outcomes, and fetal outcomes in patients diagnosed with gestational diabetes. Currently, there is very limited data on whether RT-CGM use helps patients diagnosed with gestational diabetes. By conducting this study, the investigator hopes to develop a deeper understanding of how use of a RT-CGM may affect glucose control in the gestational diabetes population.

DETAILED DESCRIPTION:
Pregnant Participants diagnosed with gestational diabetes are being invited to take part in a research study because these participants are pregnant and have gestational diabetes. Participants will be offered an opportunity to wear a medical device that monitors blood sugars (glucose). This device is called a continuous glucose monitor (CGM). The CGM measures glucose levels through a tiny plastic filament that is inserted under the skin in the abdomen by a skin prick. Typically, participants cannot feel this device once it is inserted. If participants agree to participate in this study, participants will be randomly placed into one of two groups: (1) the intervention group or (2) the control group. Participants will have a 50% (1 out of 2) chance like a coin toss of being placed into either group. If participants are in the intervention group, they will wear a real-time continuous glucose monitoring device (RT-CGM). The RT-CGM will allow participants to see glucose levels in real time. The RT-CGM will send information about glucose levels to a phone or display device so participants may see the glucose at all times. If participants are in the control group, they will not be given a RT-CGM. Instead, participants will be given a blinded CGM device. You will not be able to view your blood sugar results on the blinded CGM device. If participants are in the control group, they will also be given a blood glucose meter to check glucose using finger sticks according to the recommendations of the provider.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnancy and Gestation < 30 weeks
2. Singleton pregnancy
3. Confirmed gestational diabetes (by 75g or 100g oral glucose tolerance test or HbA1c)
4. Able to read English and completed 6th grade
5. Is able to read, understand, and sign the Informed Consent Form (ICF) and if applicable, an Authorization to Use and Disclose Protected Health Information form (consistent with Health Insurance Portability and Accountability Act of 1996 [HIPAA] legislation), communicate with the investigator, and understand and comply with protocol requirements

Exclusion Criteria:

1. Pre-gestational Type 1 or Type 2 diabetes.
2. Newly diagnosed overt-diabetes in pregnancy [HbA1c ≥ 48 mmol/mol (6.5%), fasting glucose ≥ 7.0 mmol/l, random glucose ≥ 11.1 mmol/l].
3. Pregnancies with established fetal anomalies (aside from echogenic intracardiac foci and/or renal pyelectasis) or possible preterm delivery secondary to maternal disease besides GDM
4. Known endogenous/exogenous Cushing's syndrome
5. Known chronic infections
6. Current use of any oral form of steroid medication
7. Already receiving continuous glucose monitoring (CGM)
8. History of bariatric surgery
9. Gestational Age less than 14 weeks -

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — A female who is pregnant
Enrollment: 105 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Ehrhardt, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group Blinded CGM: If you are in the control group, you will wear a continuous glucose monitor with the read out screen covered so you can not see your continuous glucose level.
- RT CGM Intervention Group: Real time continuous glucose monitor
Period: Overall Study
Arm/Group | Control Group Blinded CGM | RT CGM Intervention Group
Started | 52 | 53
Completed | 21 | 48
Not Completed | 31 | 5
Not completed — Withdrawal by Subject | 31 | 5

BASELINE CHARACTERISTICS:
Groups:
- Blinded CGM: Blinded Continuous monitoring device
- RT- CGM: Real time Continuous monitoring device
- Total: Total of all reporting groups
Arm/Group | Blinded CGM | RT- CGM | Total
Number analyzed (Participants) | 21 | 48 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (5.1) | 34.2 (5.0) | 33.7 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 48 | 69
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 17 | 40 | 57
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 14 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 23 | 30
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Glucose
Description: mean glucose CGM
Time Frame: 36 weeks
Population: Participants with > 3 days of CGM data available at 36 weeks EGA
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Blinded Continuous Glucose Monitoring Devise: If you are in the control group, you will wear a continuous glucose monitor with the read out screen covered so you can not see your continuous glucose level. You will be taught how to test your blood sugar by pricking your finger and using a standard blood glucose meter as per the standard of care used by your provider in the obstetrics clinic.
- RT-CGM: RT-CGM device wear
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 18 | 45
mg/dl | 103.0 (10.9) | 106.2 (9.6)

2. Primary Outcome: TIR CGM
Description: Time in range, 63 - 140 mg/dL (TIR) by % continuous glucose monitoring
Time Frame: 36 weeks
Population: Participants with > 3 days of CGM data at 36 weeks EGA
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 18 | 45
% of time | 92.1 (8.5) | 92.4 (7.8)

3. Secondary Outcome: Fetal Birthweight
Description: Birth weight [grams; mean (SD)]
Time Frame: delivery
Population: fetal live births with data available from hospital record or 1 self reported
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 20 | 45
grams | 3309.5 (558) | 3198.2 (486.5)

4. Secondary Outcome: TBR CGM GDM
Description: Time below range, 63 mg/dL threshold (TBR63) GDM
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 18 | 45
% of time | 1.5 (1.9) | 0.4 (0.5)

5. Secondary Outcome: TAB CGM GDM
Description: Time above range, 140 mg/dL threshold (TAR140)
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 18 | 45
% of time | 6.4 (8.5) | 7.1 (8.0)

6. Secondary Outcome: MAGE CGM
Description: Mean Amplitude of glycemic excursions (MAGE) continuous glucoe monitoring
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 18 | 45
mg/dl | 33.9 (7.0) | 34.0 (7.7)

7. Secondary Outcome: SD CGM
Description: standard deviation Continuous glucose monitoring
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 18 | 45
mg/dl | 18.6 (4.0) | 18.8 (4.3)

8. Secondary Outcome: CV CGM
Description: Coefficient of variation, % (CV)The Coefficient of Variation (%CV) is calculated by dividing the glucose Standard Deviation by the mean glucose. The %CV is a standardized measure that assesses the magnitude of glucose variability. The larger the %CV, the larger the variability in CGM readings.
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 18 | 45
percentage of variation | 18.1 (3.5) | 17.6 (3.1)

9. Secondary Outcome: Neonatal Hypoglycemia
Description: number(%) <40mg/dl of neonatal hypoglycemia
Time Frame: delivery
Population: in livebirths with glucose available in the electronic medical record
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 19 | 41
Participants | 0 | 4

10. Secondary Outcome: Gestational Age at Delivery
Description: gestational age at delivery weeks mean (sd)
Time Frame: delivery
Population: gestational age of participants with data available
Measure: Mean (Standard Deviation); unit: total time in weeks
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 44
total time in weeks | 39.0 (1.6) | 38.5 (1.5)

11. Secondary Outcome: Mode of Delivery
Description: mode of deliver reported ( vaginal, c-section, operative vaginal)
Time Frame: delivery
Population: participants with data available for mode of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 44
Participants
  c-section | 9 | 15
  vaginal | 12 | 29
  operative vaginal | 0 | 0

12. Secondary Outcome: Type of Labor
Description: Labor Status on Admission -(induced, spontaneous, planned c-section
Time Frame: delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 44
Participants
  spontaneous | 11 | 21
  induced | 2 | 9
  planned c-section | 8 | 14

13. Secondary Outcome: Shoulder Dystocia
Description: number with shoulder dystocia at delivery
Time Frame: delivery
Population: data of participants with delivery data available
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 44
Participants | 0 | 0

14. Secondary Outcome: Preeclampsia or HTN
Description: Preeclampsia or Gestational hypertension (HTN )
Time Frame: delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 44
Participants | 2 | 7

15. Secondary Outcome: Maternal Weight Gain
Description: Maternal weight gain [lbs; mean (SD)] at delivery
Time Frame: delivery
Population: Participants with weight gain data at delivery, some missing data
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 15 | 35
pounds | 21.1 (7.8) | 18.9 (9.5)

16. Secondary Outcome: Diabetes Medication Use
Description: use of metformin and insulin in pregnancy
Time Frame: at 36 weeks
Population: all participants who completed
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 48
Participants | 2 | 10

17. Secondary Outcome: 5 Minute Apgar
Description: 5 minute apgar score A 5-minute Apgar score is a quick assessment of a newborn's overall health, particularly their ability to transition to life outside the womb. It's a score between 0 and 10, with each component (appearance, pulse, grimace, activity, and respirations) receiving a score of 0, 1, or 2. A score of 7-10 is considered reassuring, while scores below 7 may indicate the need for medical attentio
Time Frame: delivery
Population: of patient's baby's with data available at delivery some missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 44
units on a scale | 9 (0.2) | 9 (0.2)

18. Secondary Outcome: Live Birth or Stillbirth
Description: live birth or still birth at delivery
Time Frame: devlivery
Population: with EMR data available about delivery or self reported
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 48
Participants
  live | 21 | 48
  still | 0 | 0

19. Secondary Outcome: Birthweight Ratio
Description: Birthweight ratio Birth weight ratio is defined as the ratio of observed birth weight divided by the median birth weight of the population-specific reference growth curve (based on 50% weight for gestational age). It is used to compare the birth weight of a fetus to the median for its gestational age. Higher birth weight ratios indicate larger fetuses for their gestational age, while lower ratios indicate smaller fetuse.
Time Frame: delivery
Population: of participant that had birthweights available at birth and gestational age at delivery,
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Blinded Continuous Glucose Monitoring Devise: blinded cgm
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 20 | 43
ratio | 1.015 (.1332) | 0.99 (0.1097)

20. Secondary Outcome: NICU Admission
Description: Need for neonatal intensive care admission
Time Frame: delivery
Population: of data available at delivery some data missing as delivered at outside hospital without record accesss or by self-report by participant
Measure: Number; unit: participants' infant
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 19 | 45
participants' infant | 1 | 3

21. Secondary Outcome: Neonatal Complications
Description: neonatal respiratory distress, birth injury, hypoxic encephalopathy
Time Frame: delivery
Population: fetal data available on EMR review some data not available as delivered outside source
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 19 | 45
Participants
  respiratory distress | 1 | 1
  birth injury | 0 | 0
  hypoxic encephalopathy | 0 | 0
  none | 18 | 44

22. Secondary Outcome: Glucose Meter Fingerstick Per Day
Description: mean number of fingersticks per day by 36 weeks
Time Frame: 36 weeks
Population: participants with fingerstick data available at 36 weeks EGA ; some missing data as participants did not provide glucose meter data
Measure: Mean (Standard Deviation); unit: fingersticks per day
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 14 | 17
fingersticks per day | 3.4 (0.8) | 0.9 (1.0)

23. Secondary Outcome: Mean Days of RT-CGM Use
Description: Mean (SD) days of RT-CGM use
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: days worn
Groups:
- RT_CGM Group: RT-CGM device use
Arm/Group | RT_CGM Group
Number analyzed (Participants) | 47
days worn | 64.4 (19.4)

24. Secondary Outcome: A1c
Description: A1c at 36 weeks
Time Frame: 36 weeks
Population: participants with A1c at 36 weeks some missing data
Measure: Mean (Standard Deviation); unit: % of A1c
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 18 | 37
% of A1c | 5.4 (0.4) | 5.4 (0.4)

25. Secondary Outcome: Fructosamine
Description: frucosamine at 36 weeks
Time Frame: 36 weeks
Population: participants with fructoasmine data at 36 weeks Some missing data
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 16 | 37
umol/L | 191.9 (11.4) | 194.7 (20.1)

26. Secondary Outcome: Short Food Questionnaire
Description: starting the conversation food questionnaire Possible scores range from 0 to 16 with lower scores indicating better nutrition including more fruits and vegtables, and less or no sugared beverages.. The most healthful answer for each question is scored 0. The less healthful answer is scored 1. The least healthful answer is scored 2.
  To get a total score, add up the individual item scores. The total score ranges from 0 to 16.
  Lower scores indicate better nutrition
Time Frame: 36 weeks
Population: of those that answered the short food question survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group Blinded CGM | RT CGM Intervention Group
Number analyzed (Participants) | 21 | 48
score on a scale | 3.8 (1.8) | 5.7 (1.8)

27. Secondary Outcome: WHO QOL Scale
Description: World health organization Quality of Life survey Possible scores range from 0 to 25 with higher scores indicating more happiness or contentment.
Time Frame: 36 weeks
Population: of those that answered the QOL survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group Blinded CGM | RT CGM Intervention Group
Number analyzed (Participants) | 18 | 45
units on a scale | 16.2 (3.6) | 15.3 (3.6)

28. Secondary Outcome: Diabetes Distress(PAID) Survey
Description: 5 items diabetes distress score Possible total score ranges from 0 to 20. Higher scores indicate more emotional distress.
Time Frame: 36 weeks
Population: of those that answered the paid survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group Blinded CGM | RT CGM Intervention Group
Number analyzed (Participants) | 21 | 48
score on a scale | 7.0 (4.9) | 8.9 (4.9)

29. Secondary Outcome: Walking Time Physcial Active Questionnaire
Description: % of participants walking greater than 10 minutes or more per day
Time Frame: 36 weeks
Population: over those that answered the physical activity survey
Measure: Number; unit: percentage of participants
Arm/Group | Control Group Blinded CGM | RT CGM Intervention Group
Number analyzed (Participants) | 21 | 45
percentage of participants | 95 | 100

30. Secondary Outcome: Metformin Only Use
Description: use of metformin only
Time Frame: at 36 weeks
Population: all participants who completed
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 48
Participants | 4 | 8

31. Secondary Outcome: Insulin Use Only
Description: use of insulin only
Time Frame: at 36 weeks
Population: all participants who completed
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 48
Participants | 1 | 14

32. Secondary Outcome: Insulin Use Only
Description: use of insulin only
Time Frame: at delivery
Population: all participants who completed
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 48
Participants | 1 | 14

33. Secondary Outcome: Diabetes Medication Use Delivery
Description: use of metformin and insulin in pregnancy
Time Frame: at delivery
Population: all participants who completed
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 48
Participants | 2 | 11

34. Secondary Outcome: Metformin Use Only at Delivery
Description: use of metformin only at time of delivery
Time Frame: at delivery
Population: all participants who completed
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Continuous Glucose Monitoring Devise | RT-CGM
Number analyzed (Participants) | 21 | 48
Participants | 3 | 7

ADVERSE EVENTS:
Time Frame: 3 to 6.5 months(duration of pregnancy)
Arm/Group | Blinded CGM | RT- CGM
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/48
Other Adverse Events (participants affected / at risk) | 0/21 | 3/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded CGM (N=21) | RT- CGM (N=48)
bleeding or irritation at device site (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) — minor bleeding or irritation at device site

LIMITATIONS AND CAVEATS:
high dropout rate/withdrawal immediately after randomization leading to lower number of subject analysis. Unreliable data given reporting in EMR varied for certain metrics for maternal/fetal outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04803357/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT04803357/ICF_001.pdf